CLINICAL TRIAL: NCT02115230
Title: Transcatheter Renal Denervation in Heart Failure With Normal Left Ventricular Ejection Fraction - a Safety and Efficacy Study of Irrigated Radiofrequency Catheter
Brief Title: Renal Denervation in Patients With Heart Failure With Normal LV Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Pedro A. Lemos, Pedro A. Lemos, Professor of Medicine, InCor Heart Institute, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IncorRDN-ICFEN
Record Dates: First submitted 2014-04-13; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Heart Failure, Diastolic; Hypertension
Keywords: Heart Failure; Heart Failure, Diastolic; Hypertension; Renal Denervation; Irrigated Radiofrequency Catheter
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal denervation + medical therapy (Experimental): Renal sympathetic denervation with an irrigated radiofrequency catheter with Celsius Thermocool (Biosense Webster, California, USA) + standard optimized medical therapy for diastolic heart failure
  Interventions: Procedure: Renal denervation + medical therapy
- Medical therapy (No Intervention): Standard optimized medical therapy for diastolic heart failure

INTERVENTIONS:
Procedure: Renal denervation + medical therapy — Renal denervation + medical therapy Renal sympathetic denervation with an irrigated radiofrequency catheter with Celsius Thermocool (Biosense Webster, California, USA) + standard optimized medical therapy for diastolic heart failure
  Arms: Renal denervation + medical therapy

SUMMARY:
It is a randomized prospective controlled study of transcatheter renal denervation in patients with Heart Failure With Normal LV Ejection Fraction. The purpose of the study is to evaluate the safety and effectiveness of renal denervation in patients with Heart Failure With Normal LV Ejection Fraction, due to reduction in renal and systemic sympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension treated with at least 2 antihypertensive drugs;
* Heart failure with a normal LV ejection fraction;
* Left Ventricular Hypertrophy (LV mass index > 96 g/m2 in women and > 116 g/m2 in men);
* ≥ 18 years of age;

Exclusion Criteria:

* Known secondary cause of hypertension
* Uncontrolled blood pressure (≥ 180x110mmHg)
* Unsuitable anatomy of renal arteries, renal stenosis or previous treatment with balloon or stent
* Advanced renal insufficiency (estimated glomerular filtration rate (GFR) < 30 ml/min/1.73 square meters)
* Diabetes Mellitus type 1
* Acute coronary syndrome or a cerebrovascular accident in the last 6 months
* Known other cause of respiratory dysfunction
* Previous LV systolic dysfunction (LVEF < 50%)
* Restrictive cardiomyopathy or Hypertrophic cardiomyopathy
* Significant valvar dysfunction
* Atrial flutter or atrial fibrillation
* Use of the oral anticoagulants
* Drug and Alcohol dependence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Change from baseline E/E' on echocardiography at 12 months | 12 months after treatment
Safety: Composite of death, myocardial infarction, cerebrovascular event, need of intervention on renal arteries and renal function impairment (decrease in estimated GFR > 30% from baseline) | 12 months

SECONDARY OUTCOMES:
Change from baseline E/E' on echocardiography at 6 months | 6 months
Change of office blood pressure and ambulatory blood pressure monitoring (ABPM) between baseline and 12 months | 12 months
Change in any echocardiographic diastolic parameter between baseline and 12 months | 12 months
Change in 6 min walking distance between baseline and 12 months | 12 months
Change in quality of life (Minnesota Living with Heart Failure Questionnaire) between baseline and 12 months | 12 months
Change in serum B-type natriuretic peptide (BNP) between baseline and 12 months | 12 months
Change in peripheral sympathetic activity measured by microneurography between baseline and 12 months | 12 months
Change in non-invasive hemodynamic parameters provided by Finometer between baseline and 12 months | 12 months
Change in renal function (GFR, albuminury and 24h urinary Na excretion) between baseline and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A Lemos, MD PhD, Study Chair — Heart Institute - InCor. University of Sao Paulo Medical School
Locations (1):
- Heart Institute - InCor. University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil